CLINICAL TRIAL: NCT00188006
Title: Biocompatible Cardiopulmonary Bypass and Neuropsychological Outcome After Coronary Artery Bypass Surgery
Brief Title: Complement Activation and Central Nervous System Injury After Coronary Artery Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PL 97-01
Record Dates: First submitted 2005-09-09; First posted 2005-09-16 (Estimated); Last update posted 2005-09-16 (Estimated); Status verified 2005-09

CONDITIONS: Coronary Artery Bypass Grafting
Keywords: cardiopulmonary bypass, inflammatory response; neurologic injury; neurocognitive deficit; biomaterials; coronary artery bypass surgery

INTERVENTIONS:
Device: heparin-coated cardiopulmonary bypass

SUMMARY:
The impact of the postoperative inflammatory response on the central nervous system after cardiac surgery is uncertain.

The goal of this study was to evaluate the role of complement activation on cellular brain injury and neurological functioning in patients undergoing coronary artery surgery. In addition, the effect of complement activation on the cerebral vasomotricity was assessed.

Because receptors to activated complement are present on astrocytes, the heparin-coated cardiopulmonary bypass that reduces complement activation should minimize these postoperative neurological adverse events. Heparin-coating might also influence blood flow velocity in cerebral arteries postoperatively if complement activation mediates cardiopulmonary bypass induced cerebral vasomotor dysfunction.

DETAILED DESCRIPTION:
Closed cardiopulmonary bypass and controlled suctions of pericardial shed blood were standardized in all patients.

Bedside transcranial Doppler examination served to evaluate the development of cerebral vasomotor dysfunction in a subgroup of patients.

ELIGIBILITY:
Inclusion Criteria:

* men undergoing coronary artery bypass surgery using cardiopulmonary bypass

Exclusion Criteria:

* clinical conditions expected to potentially influence the magnitude of the systemic inflammatory response after surgery such as open heart surgery, women because they show higher complement activation after surgery, redo cases, organ dysfunction as defined by the Euroscore such as chronic airway disease or renal dysfunction with creatinine level above 200 µmol/L, patients with left ventricular ejection fraction below 35%, diabetes mellitus under insulin therapy prior to the operation, presence of active inflammatory disease or patients taking anti-inflammatory drugs (except acetylsalicylic acid).
* significant carotid artery stenoses (>70%) at the preoperative echo-doppler examination, evidence of preexisting neurologic or psychiatric disease, existence of preoperative neuropsychological impairment as defined by preoperative Mini-Mental State Examination (MMSE) below 27, and alcohol addiction.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult

PRIMARY OUTCOMES:
sC5b-9 release
s100beta release

SECONDARY OUTCOMES:
changes in neuropsychological functioning (z scores of cognitive domains)
blood flow velocity in the middle cerebral artery (subgroup)

CONTACTS AND LOCATIONS:
Overall Officials: Christophe BAUFRETON, MD PhD, Principal Investigator — University Hospital of Angers, France

REFERENCES:
- [Result] Baufreton C, Allain P, Chevailler A, Etcharry-Bouyx F, Corbeau JJ, Legall D, de Brux JL. Brain injury and neuropsychological outcome after coronary artery surgery are affected by complement activation. Ann Thorac Surg. 2005 May;79(5):1597-605. doi: 10.1016/j.athoracsur.2004.08.061. PMID 15854939
- See also: The CardioThoracic Surgery Network — http://www.ctsnet.org/home/cbaufreton
- See also: University Hospital of Angers, France — http://www.chu-angers.fr/